CLINICAL TRIAL: NCT07173062
Title: Algae Effects in Markers of Cardiovascular Risk and Gut Microbiome: a Placebo-controlled Randomized Double-blind Trial
Brief Title: Algae Effects in Markers of Cardiovascular Risk and Gut Microbiome
Acronym: CALGUT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Centro Hospitalar De São João, E.P.E. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CALGUT
Record Dates: First submitted 2025-08-12; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Stroke; Coronary Arterial Disease (CAD); Myocardial Infarction (MI); Diabetes Mellitus; Peripheral Artery Disease (PAD); Chronic Kidney Disease(CKD); Albuminuria
Keywords: Spirulina Arthrospira platensis; Gelidium corneum; Trimethylamine- N-oxide (TMAO); Short-Chain Fatty Acids (SCFA); Cardiovascular risk (CVR)
MeSH Terms: conditions — Stroke; Myocardial Infarction; Diabetes Mellitus; Peripheral Arterial Disease; Renal Insufficiency, Chronic; Albuminuria

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double-blind, two-treatment, one-period, parallel trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Spirulina Arthrospira platensis (Experimental): during 20 weeks
  Interventions: Dietary Supplement: Spirulina Arthrospira platensis (microalgae)
- Gelidium corneum (Experimental): during 20 weeks
  Interventions: Dietary Supplement: Gelidium corneum
- Placebo (Placebo Comparator): during 20 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Spirulina Arthrospira platensis (microalgae) — Spirulina Arthrospira platensis (4 x ~500mg), taken twice daily as 2 capsules in the morning + 2 capsules in the evening
  Arms: Spirulina Arthrospira platensis
Dietary Supplement: Gelidium corneum — Gelidium corneum (4 x ~500mg), taken twice daily as 2 capsules in the morning + 2 capsules in the evening
  Arms: Gelidium corneum
Other: Placebo — Microcrystalline cellulose, silicon dioxide and dicalcium phosphate (4 x ~500mg), taken twice daily as 2 capsules in the morning + 2 capsules in the evening
  Arms: Placebo

SUMMARY:
The Western diet, rich in fat and sugar, contributes to cardiovascular risk and alters the body metabolism, specifically through the modulation of the microbiome. Microbiome is considered the "second genome", functioning as an endocrine-like organ. Gut microbiota-derived metabolites, namely trimethylamine- N-oxide and short-chain fatty acids have been associated with atherosclerosis, vascular and cardiac diseases. Regarding trimethylamine- N-oxide, its association with cardiovascular disease is positive and dose-dependent. In contrast, short-chain fatty acids have been positively associated with the improvement of cardiovascular health.

Algae probiotics can modulate gut microbiome, stimulating the growth of commensal micro-organisms with health benefits. Previous studies suggested that Spirulina Arthrospira platensis supplementation could improve blood lipid levels and lower blood pressure, revealing anti-inflammatory and antioxidant roles. Other probiotics that could be beneficial to gut microbiota are macroalgae or seaweed. Macroalgae are a rich source of components which may prompt bacterial diversity and abundance.

The present prospective, randomized, three-armed parallel trial aims to generate good-quality evidence about the potential health effects and impact of Spirulina Arthrospira platensis (microalgae) and Gelidium corneum (macroalgae) supplements in humans. These participants will undergo 3 clinical evaluations: 2 before the beginning of micro- and macro-algae supplementation and the last one after 20 weeks of supplementation. The evaluation includes a vascular, nutritional and physical activity assessment, as well as blood, urine, saliva and stool collection for quantification of plasma biomarkers, oral and gut microbiota analysis, respectively.

ELIGIBILITY:
Inclusion Criteria:

* ≥50 years
* BMI ≥20 kg/m2
* History of stroke, coronary artery disease, myocardial infarction, peripheral artery disease, chronic kidney disease (eGFR <75 ml/min at least for 3 months), albuminuria >300 mg/g, or diabetes mellitus
* No antibiotics in the previous 30 days
* If a woman, she must be a woman of non-childbearing potential. That is, she must be:

  * Surgically sterilized (e.g. underwent hysterectomy, bilateral salpingectomy or bilateral oophorectomy);
  * Clinically diagnosed infertile;
  * In a post-menopausal state, defined as no menses for 12 months without an alternative medical cause.
* A woman patient of childbearing potential must have a negative serum pregnancy test at Visit 0 (Day 0) and must agree to use consistently and correctly (from 28 days prior to first study treatment administration until at least 7 days after last study treatment administration) one of the following highly effective methods of contraception:

  * Abstinence of heterosexual intercourse (when this is in line with preferred and usual lifestyle of the subject);
  * Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable);
  * Combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal);
  * Intrauterine device;
  * Intrauterine hormone-releasing system;
  * Bilateral tubal occlusion;
  * Vasectomized partner, who has received medical assessment of the surgical success, or clinically diagnosed infertile partner.

Exclusion Criteria:

* Unwilling to sign the informed consent form (if the patient wants to participate but cannot sign for any reason, then a third-person testimony may sign/complete the informed consent form on the patient's behalf).
* Involvement in the planning and/or conduct of the study (applies to both Investigator staff and/or staff at the study site).
* Participation in another clinical study with an investigational product during the last month.
* In participants recruited at Unidade Local de Saúde de São João, the exclusion criteria applied is estimated Glomerular Filtration Rate (eGFR) <30 ml/min/1.73m2 estimated with the CKD-EPI (2021) formula or dialysis. For participants recruited at community, this exclusion criteria is adapted for diagnosis of end-stage renal disease or dialysis (no need to quantify the eGFR).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Plasma trimethylamine-N-oxide levels | Visit 1 (day 7 to day 30) and Visit 2 (20 weeks ± 15 days from Visit 1)
  To assess the effect of the Spirulina Arthrospira platensis versus Gelidium corneum versus placebo on the between-group ratio of geometric means difference of the Log transformed plasma trimethylamine- N-oxide levels change from baseline to 20 weeks.
  The co-primary comparison will be Spirulina Arthrospira platensis versus Placebo and Gelidium corneum versus Placebo with a 2.5% alfa for each comparison.

SECONDARY OUTCOMES:
Plasma short-chain fatty acids levels | Visit 1 (day 7 to day 30) and Visit 2 (20 weeks ± 15 days from Visit 1)
  To assess the effect of the Spirulina Arthrospira platensis versus Gelidium corneum versus placebo on the percentage change of the following measures relative to the baseline measures.
Gut microbiota | Visit 1 (day 7 to day 30) and Visit 2 (20 weeks ± 15 days from Visit 1)
  To assess the effect of the Spirulina Arthospira platensis versus Gelidium corneum versus placebo on the percentage change of the following measures relative to the baseline measures.
Systolic blood pressure | Visit 1 (day 7 to day 30) and Visit 2 (20 weeks ± 15 days from Visit 1)
  To assess the effect of the Spirulina Arthrospira platensis versus Gelidium corneum versus placebo on the percentage change of the following measures relative to the baseline measures.
Diastolic blood pressure | Visit 1 (day 7 to day 30) and Visit 2 (20 weeks ± 15 days from Visit 1)
  To assess the effect of the Spirulina Arthrospira platensis versus Gelidium corneum versus placebo on the percentage change of the following measures relative to the baseline measures.
Body weight | Visit 1 (day 7 to day 30) and Visit 2 (20 weeks ± 15 days from Visit 1)
  To assess the effect of the Spirulina Arthrospira platensis versus Gelidium corneum versus placebo on the percentage change of the following measures relative to the baseline measures.
Total cholesterol | Visit 1 (day 7 to day 30) and Visit 2 (20 weeks ± 15 days from Visit 1)
  To assess the effect of the Spirulina Arthrospira platensis versus Gelidium corneum versus placebo on the percentage change of the following measures relative to the baseline measures.
Low-density lipoprotein cholesterol | Visit 1 (day 7 to day 30) and Visit 2 (20 weeks ± 15 days from Visit 1)
  To assess the effect of the Spirulina Arthrospira platensis versus Gelidium corneum versus placebo on the percentage change of the following measures relative to the baseline measures.
High-density lipoprotein cholesterol | Visit 1 (day 7 to day 30) and Visit 2 (20 weeks ± 15 days from Visit 1)
  To assess the effect of the Spirulina Arthrospira platensis versus Gelidium corneum versus placebo on the percentage change of the following measures relative to the baseline measures.
Lipoprotein A | Visit 1 (day 7 to day 30) and Visit 2 (20 weeks ± 15 days from Visit 1)
  To assess the effect of the Spirulina Arthrospira platensis versus Gelidium corneum versus placebo on the percentage change of the following measures relative to the baseline measures.
Triglycerides | Visit 1 (day 7 to day 30) and Visit 2 (20 weeks ± 15 days from Visit 1)
  To assess the effect of the Spirulina Arthrospira platensis versus Gelidium corneum versus placebo on the percentage change of the following measures relative to the baseline measures.
Interleukin-6 | Visit 1 (day 7 to day 30) and Visit 2 (20 weeks ± 15 days from Visit 1)
  To assess the effect of the Spirulina Arthrospira platensis versus Gelidium corneum versus placebo on the percentage change of the following measures relative to the baseline measures.
Glucose | Visit 1 (day 7 to day 30) and Visit 2 (20 weeks ± 15 days from Visit 1)
  To assess the effect of the Spirulina Arthrospira platensis versus Gelidium corneum versus placebo on the percentage change of the following measures relative to the baseline measures.
Insulin | Visit 1 (day 7 to day 30) and Visit 2 (20 weeks ± 15 days from Visit 1)
  To assess the effect of the Spirulina Arthrospira platensis versus Gelidium corneum versus placebo on the percentage change of the following measures relative to the baseline measures.
Haemoglobin A1c | Visit 1 (day 7 to day 30) and Visit 2 (20 weeks ± 15 days from Visit 1)
  To assess the effect of the Spirulina Arthrospira platensis versus Gelidium corneum versus placebo on the percentage change of the following measures relative to the baseline measures.
Estimated Glomerular Filtration Rate | Visit 1 (day 7 to day 30) and Visit 2 (20 weeks ± 15 days from Visit 1)
  To assess the effect of the Spirulina Arthrospira platensis versus Gelidium corneum versus placebo on the percentage change of the following measures relative to the baseline measures.
Sodium | Visit 1 (day 7 to day 30) and Visit 2 (20 weeks ± 15 days from Visit 1)
  To assess the effect of the Spirulina Arthrospira platensis versus Gelidium corneum versus placebo on the percentage change of the following measures relative to the baseline measures.
Potassium | Visit 1 (day 7 to day 30) and Visit 2 (20 weeks ± 15 days from Visit 1)
  To assess the effect of the Spirulina Arthrospira platensis versus Gelidium corneum versus placebo on the percentage change of the following measures relative to the baseline measures.
High-sensitivity C-reactive protein | Visit 1 (day 7 to day 30) and Visit 2 (20 weeks ± 15 days from Visit 1)
  To assess the effect of the Spirulina Arthrospira platensis versus Gelidium corneum versus placebo on the percentage change of the following measures relative to the baseline measures.
Oral microbiota | Visit 1 (day 7 to day 30) and Visit 2 (20 weeks ± 15 days from Visit 1)
  To assess the effect of the Spirulina Arthrospira platensis versus Gelidium corneum versus placebo on the percentage change of the oral microbiota relative to the baseline.
Pulse wave velocity | Visit 1 (day 7 to day 30) and Visit 2 (20 weeks ± 15 days from Visit 1)
  To assess the effect of the Spirulina Arthrospira platensis versus Gelidium corneum versus placebo on arterial stiffness.
  Measured by carotid-femoral pulse wave velocity using pulse wave analysis to assess arterial stiffness. Expressed in m/s. Higher values = greater arterial stiffness.
Intima-media thickness | Visit 1 (day 7 to day 30) and Visit 2 (20 weeks ± 15 days from Visit 1)
  To assess the effect of Spirulina Arthrospira platensis versus Gelidium corneum versus placebo on vascular structure, measured by carotid intima-media thickness using cervical echo-Doppler ultrasound.
  Measured by cervical echo-Doppler ultrasound in the common carotid artery (automatic recording of 5 cycles). Expressed in mm. Lower values = better vascular structure.
Cerebral blood flow velocities | Visit 1 (day 7 to day 30) and Visit 2 (20 weeks ± 15 days from Visit 1)
  To assess the effect of the Spirulina Arthrospira platensis versus Gelidium corneum versus placebo on cerebral blood flow.
  Measured by transcranial color-coded duplex Doppler in middle cerebral arteries and posterior cerebral arteries. Expressed in cm/s. Higher values = greater blood flow velocity.
Cerebral blood flow resistance indexes | Visit 1 (day 7 to day 30) and Visit 2 (20 weeks ± 15 days from Visit 1)
  To assess the effect of the Spirulina Arthrospira platensis versus Gelidium corneum versus placebo on cerebral vascular resistance.
  Measured by transcranial color-coded duplex Doppler in middle cerebral arteries and posterior cerebral arteries. Expressed as resistance index (RI), calculated from Doppler waveforms. Higher RI = greater vascular resistance.
Cerebral vascular reactivity | Visit 1 (day 7 to day 30) and Visit 2 (20 weeks ± 15 days from Visit 1)
  To assess the effect of the Spirulina Arthrospira platensis versus Gelidium corneum versus placebo on cerebral vascular reactivity.
  Measured by transcranial color-coded duplex Doppler during a breathing manoeuvre. Expressed as % change in blood flow velocity in middle cerebral arteries and posterior cerebral arteries, in response to hypercapnia. Greater reactivity = better cerebrovascular function.
Breath-holding index | Visit 1 (day 7 to day 30) and Visit 2 (20 weeks ± 15 days from Visit 1)
  To assess the effect of the Spirulina Arthrospira platensis versus Gelidium corneum versus placebo on cerebrovascular reserve capacity.
  Measured by transcranial color-coded duplex Doppler in middle cerebral arteries and posterior cerebral arteries during a 20-second apnea manoeuvre. Expressed as index value. Higher BHI = better vascular reserve.
Neurovascular coupling (visual stimulation) | Visit 1 (day 7 to day 30) and Visit 2 (20 weeks ± 15 days from Visit 1)
  To assess the effect of the Spirulina Arthrospira platensis versus Gelidium corneum versus placebo on neurovascular coupling.
  Measured by transcranial color-coded duplex Doppler during visual stimulation with a flickering checkerboard (10 Hz). Expressed as blood velocity change in middle cerebral arteries and posterior cerebral arteries recorded across cycles of 20 seconds stimulation (eyes open) and 20 seconds rest (eyes closed). Greater change = better neurovascular coupling.
Mediterranean diet adherence screener score | Visit 1 (day 7 to day 30) and Visit 2 (20 weeks ± 15 days from Visit 1)
  To assess the effect of Spirulina Arthrospira platensis versus Gelidium corneum versus placebo on the percentage change in adherence to the Mediterranean diet, as measured by the Mediterranean Diet Adherence Screener (MEDAS).
  The MEDAS is a 14-item questionnaire that evaluates food intake habits and frequency of consumption of specific foods. Each item receives 1 point for a positive response, resulting in a total score ranging from 0 to 14. Higher scores indicate greater adherence to the Mediterranean diet, with a score of ≥10 considered adherent.
Total score of physical activity | Visit 1 (day 7 to day 30) and Visit 2 (20 weeks ± 15 days from Visit 1)
  To assess the effect of Spirulina Arthrospira platensis versus Gelidium corneum versus placebo on the percentage change in total physical activity score, as measured by the International Physical Activity Questionnaire - short version.
  This questionnaire includes 7 items assessing frequency and duration of physical activity during the past 7 days across different domains. Activities are weighted by metabolic equivalents (METs) (walking = 3, moderate = 4, vigorous = 8), and a total score is expressed as MET-minutes/week. Scores range from 0 to several thousand, with higher values indicating greater physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: João Pedro Ferreira, MD, PhD, Principal Investigator — Universidade do Porto
Locations (1):
- Unidade Local de Saúde de São João, Porto, Portugal